CLINICAL TRIAL: NCT05669040
Title: mHealth to Improve the Experience, Adherence to Drug Treatment and Positive Mental Health of Patients Diagnosed With Femur Fracture: Protocol for a Quasi-experimental Study
Brief Title: mHealth to Improve the Experience, Adherence to Drug Treatment and Positive Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Amgen (Industry); University of Barcelona (Other)
Responsible Party: Principal Investigator, Gemma Marcos, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Intervention EFE
Record Dates: First submitted 2022-12-02; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Fracture of Femur
Keywords: education; patient experience; adherence medication; mental health; mobile health; nurse; mHealth; protocol
MeSH Terms: conditions — Femoral Fractures; Medication Adherence; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient experience (Active Comparator)
  Interventions: Other: Pharmacological education; Other: Training in the use of MyPlan Aplication; Other: Patient Experience
- Adherence to drug treatment (Active Comparator)
  Interventions: Other: Pharmacological education; Other: Training in the use of MyPlan Aplication
- Positive mental health (Active Comparator)
  Interventions: Other: Patient Experience

INTERVENTIONS:
Other: Pharmacological education — Inform the patient of the medication that is being taken and how it has to be taken; What is it for and the side effects and/or adverse reactions.
  Arms: Adherence to drug treatment; Patient experience
Other: Training in the use of MyPlan Aplication — Review of the use of the aplication
  Arms: Adherence to drug treatment; Patient experience
Other: Patient Experience — * How do you feel?
  * Sad feelings and frustration.
  * Achievements day by day, think positive.
  * Importance of interpersonal relationships.
  * Explain activities to relax the mind
  Arms: Patient experience; Positive mental health

SUMMARY:
The present study aims to evaluate the effectiveness of a pharmacological nursing educational intervention (EFE) with "Myplan Aplication" about the patient's experience, adherence to pharmacological treatment, and positive mental health of patients with femur fracture.

DETAILED DESCRIPTION:
Once the informed consent has been obtained, the investigators will explain to the patient the pharmacological treatment with the support of an aplication (what it is for, how the medication should be taken, possible adverse effects), also the investigators will share time with the patient during the 4 face-to-face training sessions. The investigators will accompany during their hospital stay, offering to pacients telematic support upon discharge with the treatment and until the end of the study. This is a quasi-experimental non-randomized study with 3 phases of data collection. Possible adverse reactions, if any, will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of femur fracture
* knowledge of the Spanish language
* 24-hour admission to the traumatology unit
* level of consciousness on the Glasgow scale of 15
* have access to a mobile device
* ability to participate in the pilot study
* be able to provide written informed consent or obtain consent from a legal representative.

Exclusion Criteria:

* presence of psychological pathologies or cognitive impairment
* isolation in hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Patient experience questionnaire-15. Changes in outcomes are assessed at three time points. | at 1rst day (before intervention), at 7th day (at discharge after intervention), and 25th day (after discharge)
  This questionnaire allows us to explore the perception of patients about the information process and participation in decision-making during hospital admission. The responses range is from always or almost always/quite frequently/sometimes/never or almost never.This questionnaire allows us to explore the perception of patients about the information process and participation in decision-making during hospital admission. The responses range from always or almost always/quite frequently/sometimes/never or almost never.
Morinski-Green Questionnaire. Changes in outcomes are assessed at three time points. | at 1rst day, at 7th day and 25th day.
  This questionnaire allows assessing adherence to the prescribed treatment. It consists of a series of 4 dichotomous yes/no questions that reflects the degree of behavior of the patient's compliance, information on the causes of non-compliance.
Positive Mental Health Questionnaire. Changes in outcomes are assessed at three time points. | at 1rst day, at 7th day and 25th day.
  This scale evaluates mental health from a positive perspective. It consists of 39 items distributed in six factors: personal satisfaction, pro-social attitude, self-control, autonomy, problem solving and self-acting, and interpersonal relationship skills. Its measurement is carried out by means of a Likert-type response that goes from always or almost always, quite frequently, sometimes, never or almost never. Validated in the general population in favorable psychometric values: global reliability of 0.88 and an applied variance of 45%.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Moreno Arroyo, Study Director — UB
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
* Publication of an article with preliminary results in the BioMed Central Public Health magazine.
  * Presentation of results at National Congress of Mental Health Nursing. Spain.
  * Publication of results article in "Revista Española de Enfermería de Salud Mental" magazine.
  * Presentation of results at Investen, Annual Meeting on Care Research. Spain.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: February 2024
Access Criteria: Healthcare professionals